CLINICAL TRIAL: NCT05442034
Title: Rh-PDGF Versus Emdogain for Treatment of Intra-bony Defects
Brief Title: Rh-PDGF vs EMD for Treatment of Intra-bony Defects
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-217-NSU
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Intrabony Periodontal Defect
Keywords: Periodontal regeneration; Inta-bony defects; Enamel matrix derivatives
MeSH Terms: interventions — Regeneration

STUDY DESIGN:
Intervention Model Description: Test group will receive rh-PDGF in combination with bone allograft Control group will receive EMD in combination with bone allograft.
Who Masked: Participant
Masking Description: Participants will not know which biologic agent (rh-PDGF or EMD) is being used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- recombinant human platelet derived growth factor (rh-PDGF) in combination with bone allograft (Experimental): recombinant human platelet derived growth factor is a protein that is found in blood serum. It helps to recruit stem cells into the area to aid in cell differentiation and proliferation. When added to mineralized bone allograft, it stimulates the angiogenesis in the area, and this in turn may increase the outcomes of regeneration.
  Interventions: Biological: growth factors to help in regeneration
- Enamel matrix derivatives (EMD) in combination with bone allograft. (Active Comparator): Enamel matrix derivatives are natural proteins that are produced in the developing dental follicle. It has been available for decades and has been proved to help in regeneration of intrabony defects when applied into the root surface. When combined with bone allograft, it results in regeneration of intrabony defects.
  Interventions: Biological: growth factors to help in regeneration

INTERVENTIONS:
Biological: growth factors to help in regeneration — regenerative therapy

SUMMARY:
Treatment of intra-bony defects is challenging and requires extensive knowledge of the etiology, anatomy, occlusion, and available biomaterials that can be used to treat this kind of defects. Patients who received scaling and root planing at the college of dental medicine due to periodontal disease, will be screened for inclusion. Only subjects who showed persistent deep probing depth associated with an intrabony defect will be included and will be randomly allocated to one of two treatment groups. One group will be treated using recombinant human platelet derived growth factor (GEM-21) (test) added to allogenic bone graft, second group will be treated using enamel matrix derivatives (EMD) (control) with allograft. Both groups will be treated using the same surgical protocol. Patients will be followed up for a period of 6 months, before getting re-evaluated for assessing the effectiveness of the applied therapies.

DETAILED DESCRIPTION:
Alveolar bone crest is considered normal when it is found at a distance of 0.4- 1.97mm from the cementoenamel junction (CEJ) of the tooth. Chronic inflammation resulting from periodontal disease (PD) may lead to change in this architecture and formation of osseous defects. The variation in the form of these defects may be influenced by the occlusal stresses that the tooth is subjected to or the original form of the alveolar process in a localized area.

While Glickman chose to classify the osseous defects into "Osseous craters, intra-bony defects, bulbous osseous contours, hemi-septa, inconsistent margins and ledges"; Pritchard classified them as "interproximal craters, inconsistent margins, hemi-septa, furca invasions, intra-bony defects and a combination of these defects". Identifying the type of defect is of utmost importance. Intra-bony defects found in the interproximal areas can be one-wall, two-walls, or three-walls defects, depending on how many walls are remaining. On the other hand, when the inter-radicular bone is lost, its commonly classified as grade I, grade II, or grade III furcation.

Successful regeneration of the intra-bony defects will be accompanied by clinical attachment gain, decreased pocket depth, radiographic bone height gain, and improved periodontal health, to reach this goal, several types of bone grafts, membranes, biologics and/or combinations, have been investigated for potential application and, they proved success over short- and long-term.

Flemming et al. 1998, tested the bone gain following open flap debridement (OFD) versus allogeneic bone graft. The group that received allogenic bone graft had higher bone gain compared to the OFD group at 6 months (2.2mm vs 1.2mm) and 3 years (2.3mm vs 1.1mm) (P <0.05). Comparable results were found when A. Sculean et al 2004, tested CAL gain when enamel matrix proteins (EMD) was used versus OFD; having 1.3mm of CAL gain at 5 years when the latter was used versus 2.9mm when the former was used (p<0.001). Eickholz et al. 2004, tested the use of bioabsorbable membrane for the treatment of intra-bony defects with guided tissue regeneration. Attachment height gain was stable at 12- and 60-months follow up (3.5mm and 2.2mm). In a case series, Kim et al. compared the clinical attachment gain in 12 pairs of intra-bony defects in 12 subjects. One side was randomly assigned to receive GTR with a bioabsorbable membrane (Polyglactin) (control), while the contralateral received non-resorbable membrane (e-PTFE) (test). Both groups yielded significant clinical attachment gain at 6 (C6 and T6) and 60 months (C60 and T60), (C6: 2.6 ± 1.4 mm; C60: 1.6 ± 1.5 mm; T6: 3.0 ± 1.7 mm; T60: 3.0 ± 0.7 mm).

Emdogain is a biologic material that consists of hydrophobic enamel matrix proteins extracted from developing embryogenic enamel of porcine origin. It was first tested on monkeys for ability to regenerate buccal dehiscence defects and resulted in complete regeneration of the defect. It was later used in conjunction with Modified Widman Flap (MWF) and compared to MWF with placebo, for the regeneration of intra-bony defects in human subjects. At 36 months, the EMD group yielded significantly higher bone gain (2.2 mm vs 1.7 mm), respectively.

Platelet derived growth factors (PDGF) is a human serum polypeptide growth factor, it is a potent mitogen for cells of mesenchymal origin (e.g., fibroblasts), it stimulates collagen synthesis, chemotaxis of fibroblasts and production of insulin-like growth factors (IGF). It has been tested both in vitro and in vivo, it has proved potential for promoting soft tissue wound repair, and when used in periodontal defects, it stimulated healing with new bone and cementum formation, and a deposition of a continuous layer of osteoblasts was noticed lining the newly formed bone.

Based on the above evidence, it is now clear that different techniques and biomaterials can be used for periodontal regeneration. It is the purpose of the current study, to investigate the effect of rh-PDGF (test) in its commercial form (GEM21) and enamel matrix derivatives in its commercial form (EMD) (control) in combination with allografts for the treatment of periodontal defects in one-wall and two-walls intra-bony defects in human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age is 18 years old and older
* Absence of relevant medical conditions
* Availability for 6-month follow-up
* Subjects who recently have received scaling and root planing due to periodontal disease
* Single-rooted and multi-rooted teeth in either the maxilla or the mandible.
* Presence of interdental periodontal pocket with PD ≥ 6 mm associated to an intra-bony component ranged from 3 to 6 mm.
* Non-contained intra-bony defects (1-wall, 2-wall intra-bony defects)
* Full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) <20% at surgery

Exclusion Criteria:

* Female patients who are pregnant or planning to be pregnant during the period of the study
* Heavy smokers (>10 cigarettes a day)
* Subjects not willing to comply to the study protocol
* Patients with uncontrolled diabetes (HbA1c >7.5)
* Patients receiving medications that may affect periodontal status in the previous 6 months (e.g., Phenytoin, Alendronate)
* Periapical lesion in the tested sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Changes | 6 months
  Change in gingival recession and pocket probing depth

CONTACTS AND LOCATIONS:
Overall Officials: Theofilos Koutouzis, DDS, MS, Study Director — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Davie, Florida, United States

IPD SHARING:
Plan to Share IPD: No